CLINICAL TRIAL: NCT03305900
Title: Lifestyle, Metabolite and Genetic Determinants of Formate Concentrations in a Cross-sectional Study of Young, Healthy Adults
Brief Title: Determinants of Formate Concentrations
Status: Completed | Type: Observational
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, John (Sean) Brosnan, Professor of Biochemistry, Memorial University of Newfoundland
Other Study IDs: 12.190 HREA
Record Dates: First submitted 2017-09-28; First posted 2017-10-10 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Healthy
Keywords: formate; one-carbon metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — Cross-sectional study requiring a single serum sample

SUMMARY:
Formate is an important metabolite, serving as a donor of one-carbon groups to the intracellular tetrahydrofolate pool. However, little is known of its circulating concentrations or of their determinants. This study seeks to define formate levels and their determinants in a young, healthy population.

Serum formate will be measured in 1701 subjects from the Trinity Student Study. The subjects, males and females, aged 18 to 28 years, were enrolled at Trinity College, Dublin. Formate levels will be compared with other one-carbon metabolites, vitamin status, potential formate precursors, genetic polymorphisms, and lifestyle factors.

ELIGIBILITY:
Inclusion Criteria:

* Trinity College Dublin students with Irish grandparents

Exclusion Criteria:

* None

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Serum formate was measured in 1701 subjects from the Trinity Student Study. The subjects, males and females, aged 18 to 28 years, were enrolled at Trinity College, Dublin
Sampling Method: Non-Probability Sample
Enrollment: 1701 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2013-11-26 (Actual); Study Completion 2013-11-26 (Actual)

PRIMARY OUTCOMES:
Formate concentrations | Single baseline measurement; cross sectional, observational study
  Formate concentrations in study population

CONTACTS AND LOCATIONS:
Overall Officials: Anne Molloy, Ph.D., Study Chair — University of Dublin, Trinity College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brosnan JT, Mills JL, Ueland PM, Shane B, Fan R, Chiu CY, Pangilinan F, Brody LC, Brosnan ME, Pongnopparat T, Molloy AM. Lifestyle, metabolite, and genetic determinants of formate concentrations in a cross-sectional study in young, healthy adults. Am J Clin Nutr. 2018 Mar 1;107(3):345-354. doi: 10.1093/ajcn/nqx065. PMID 29566195